CLINICAL TRIAL: NCT04980092
Title: Assessment of Kidney Function and Osteomuscular Status in Survivors of a Prolonged Stay in Intensive Care Unit
Brief Title: Assessment of Kidney Function and Osteomuscular Status After Critical Care
Status: Suspended | Type: Observational
Why Stopped: Enrollment difficulties
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, University of Liege
Other Study IDs: ROPS
Record Dates: First submitted 2021-07-09; First posted 2021-07-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Kidney Injury; Muscle Loss; Bone Loss
MeSH Terms: conditions — Critical Illness; Muscular Atrophy; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-ICU group: Observational foolow-up
  Interventions: Other: one-year follow-up

INTERVENTIONS:
Other: one-year follow-up — patients will be followed during the year after ICU discharge, in order to assess kidney function, and muscle and bone health

SUMMARY:
This observational study aims to assess kidney function through direct glomerular filtration rate (GFR) using iohexol clearance, compared to estimated GFR based on creatinine and cystatin C equations. Kidney function will also be evaluated through renal fibrosis biomarkers. Kidney function will be correlated to body composition, muscle turnover biomarkers, and bone micro-architecture.

DETAILED DESCRIPTION:
The investigators developed a post-ICU clinic where complications of the post-intensive care syndrome are detected. Muscle function is assessed by clinical testings, muscle strength measurement. Body composition is measured by electrical bioimpedance. Bone mass is assessed using dual-energy radiographic absorptiometry.

It is well known that ICU survivors experience a loss of muscle mass. This can lead to misinterpretation of estimated GFR based on creatinine equations.

The aim of the present study is to assess the evolution of kidney function after a prolonged stay in ICU, using GFR equations based on cystatin C, and to compare it to measured GFR using iohexol clearance.

The second aim is to explore the evolution of bone and muscle health in these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients surviving an ICU stay of at least 7 days
* patients who experienced acute kidney injury (KDIGO criteria) during ICU stay

Exclusion Criteria:

* chronic kidney injury with dedicated follow-up before ICU admission
* chronic extrarenal epuration
* kidney transplant
* allergy to iohexol
* iodinated contrast allergy
* refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: survivors of an ICU stay of at least 7 days
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
measured GFR | between day 0 and day 7 after ICU discharge
  plasma clearance of iohexol
measured GFR | at 3 months after ICU discharge
  plasma clearance of iohexol
measured GFR | at 12 months after ICU discharge
  plasma clearance of iohexol
estimated GFR | between day 0 and day 7 after ICU discharge
  cystatin C based CKD-EPI equation
estimated GFR | at 3 months after ICU discharge
  cystatin C based CKD-EPI equation
estimated GFR | at 12 months after ICU discharge
  cystatin C based CKD-EPI equation

SECONDARY OUTCOMES:
urine concentration of renal fibrose biomarkers | between day 0 and day 7 after ICU discharge
  urine measurement of TGF-β concentration
urine concentration of renal fibrose biomarkers | at 3 months after ICU discharge
  urine measurement of TGF-β concentration
urine concentration of renal fibrose biomarkers | at 12 months after ICU discharge
  urine measurement of TGF-β concentration
urine concentration of renal fibrose biomarkers | between day 0 and day 7 after ICU discharge
  urine measurement of monocyte chemoattractant protein-1 concentration
urine concentration of renal fibrose biomarkers | at 3 months after ICU discharge
  urine measurement of monocyte chemoattractant protein-1 concentration
urine concentration of renal fibrose biomarkers | at 12 months after ICU discharge
  urine measurement of monocyte chemoattractant protein-1 concentration
urine concentration of renal fibrose biomarkers | between day 0 and day 7 after ICU discharge
  urine measurement of matrix metalloproteinases concentration
urine concentration of renal fibrose biomarkers | at 3 months after ICU discharge
  urine measurement of matrix metalloproteinases concentration
urine concentration of renal fibrose biomarkers | at 12 months after ICU discharge
  urine measurement of matrix metalloproteinases concentration
urine concentration of renal fibrose biomarkers | between day 0 and day 7 after ICU discharge
  urine measurement of chemokine ligands concentration
urine concentration of renal fibrose biomarkers | at 3 months after ICU discharge
  urine measurement of chemokine ligands concentration
urine concentration of renal fibrose biomarkers | at 12 months after ICU discharge
  urine measurement of chemokine ligands concentration
urine concentration of renal fibrose biomarkers | between day 0 and day 7 after ICU discharge
  urine measurement of C-X-C motif chemokine ligand concentration
urine concentration of renal fibrose biomarkers | at 3 months after ICU discharge
  urine measurement of C-X-C motif chemokine ligand concentration
urine concentration of renal fibrose biomarkers | at 12 months after ICU discharge
  urine measurement of C-X-C motif chemokine ligand concentration
urine concentration of renal fibrose biomarkers | between day 0 and day 7 after ICU discharge
  measurement of proteinuria
urine concentration of renal fibrose biomarkers | at 3 months after ICU discharge
  measurement of proteinuria
urine concentration of renal fibrose biomarkers | at 12 months after ICU discharge
  measurement of proteinuria
blood concentration of muscle turnover markers | between day 0 and day 7 after ICU discharge
  blood measurement of myostatin concentration
blood concentration of muscle turnover markers | at 3 months after ICU discharge
  blood measurement of myostatin concentration
blood concentration of muscle turnover markers | at 12 months after ICU discharge
  blood measurement of myostatin concentration
blood concentration of muscle turnover markers | between day 0 and day 7 after ICU discharge
  blood measurement of procollagen type III N-terminal peptide (P3NP) concentration
blood concentration of muscle turnover markers | at 3 months after ICU discharge
  blood measurement of procollagen type III N-terminal peptide (P3NP) concentration
blood concentration of muscle turnover markers | at 12 months after ICU discharge
  blood measurement of procollagen type III N-terminal peptide (P3NP) concentration
blood concentration of muscle turnover markers | between day 0 and day 7 after ICU discharge
  blood measurement of insulin growth factor 1 concentration
blood concentration of muscle turnover markers | at 3 months after ICU discharge
  blood measurement of insulin growth factor 1 concentration
blood concentration of muscle turnover markers | at 12 months after ICU discharge
  blood measurement of insulin growth factor 1 concentration
bone micro-architecture | between day 0 and day 7 after ICU discharge
  high resolution peripheral quantitative computed tomography (HRpQCT) images acquisition
bone micro-architecture | at 3 months after ICU discharge
  high resolution peripheral quantitative computed tomography (HRpQCT) images acquisition
bone micro-architecture | at 12 months after ICU discharge
  high resolution peripheral quantitative computed tomography (HRpQCT) images acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Rousseau, MD, PhD, Principal Investigator — University hospital of Liège
Locations (1):
- University Hospital of Liège, Liège, Liège, Belgium